CLINICAL TRIAL: NCT00137189
Title: Resource-oriented Music Therapy for Psychiatric Patients With Low Therapy Motivation: A Randomised Controlled Trial
Brief Title: Resource-oriented Music Therapy for Psychiatric Patients With Low Therapy Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: The Research Council of Norway (Other); Helse Vest (Other); Helse Forde (Other); Nordfjord Psychiatric Centre (Other); Helse Stavanger HF (Other Government); Jæren District Psychiatric Centre (Unknown); The Wagner-Jauregg Provincial Neuropsychiatric Clinic (Individual); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-MTPSY
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Mental Disorders; Mood Disorders; Personality Disorders; Schizophrenia and Disorders With Psychotic Features
Keywords: Motivation; Music Therapy; Psychotherapy
MeSH Terms: conditions — Mental Disorders; Mood Disorders; Personality Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): See published study protocol
  Interventions: Procedure: Resource-oriented music therapy; Procedure: Standard care
- Standard care (Other): See published study protocol
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Resource-oriented music therapy
  Arms: Music therapy
Procedure: Standard care

SUMMARY:
The aim of this study is to examine whether resource-oriented music therapy helps psychiatric patients with low therapy motivation to improve negative symptoms and other health-related outcomes.

DETAILED DESCRIPTION:
Background: Previous research has shown positive effects of music therapy for people with schizophrenia and other mental disorders. In clinical practice, music therapy is often offered to psychiatric patients with low therapy motivation, but little research exists about this population. The aim of this study is to examine whether resource-oriented music therapy helps psychiatric patients with low therapy motivation to improve negative symptoms and other health-related outcomes. An additional aim of the study is to examine the mechanisms of change through music therapy.

Method: 144 adults with a non-organic mental disorder (ICD-10: F1 to F6) who have low therapy motivation and a willingness to work with music will be randomly assigned to an experimental or a control condition. All participants will receive standard care, and the experimental group will in addition be offered biweekly sessions of music therapy over a period of three months. Outcomes will be measured by a blind assessor before and 1, 3, and 9 months after randomisation.

Discussion: The findings to be expected from this study will fill an important gap in the knowledge of treatment effects for a patient group that does not easily benefit from treatment. The study's close link to clinical practice, as well as its size and comprehensiveness, will make its results well generalisable to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Non-organic mental disorder
* Low therapy motivation
* Willingness to work with music

Exclusion Criteria:

* Severe mental retardation
* Life-threatening somatic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
negative symptoms (Scale for the Assessment of Negative Symptoms [SANS]) | 1
negative symptoms (Scale for the Assessment of Negative Symptoms [SANS]) | 3 months
negative symptoms (Scale for the Assessment of Negative Symptoms [SANS]) | 9 months

SECONDARY OUTCOMES:
general symptoms | 1
general symptoms | 3 months
general symptoms | 9 months
general functioning | 1 months
general functioning | 3 months
general functioning | 9 months
clinical global impressions | 1 months
clinical global impressions | 3 months
clinical global impressions | 9 months
interest in music | 1 months
interest in music | 3 months
interest in music | 9 months
motivation for change | 1 months
motivation for change | 3 months
motivation for change | 9 months
self-efficacy | 1 months
self-efficacy | 3 months
self-efficacy | 9 months
self-esteem | 1 months
self-esteem | 3 months
self-esteem | 9 months
vitality | 1 months
vitality | 3 months
vitality | 9 months
affect regulation | 1 months
affect regulation | 3 months
affect regulation | 9 months
relational competence | 1 months
relational competence | 3 months
relational competence | 9 months
actual social relationships | 1 months
actual social relationships | 3 months
actual social relationships | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gold, PhD, Principal Investigator — Grieg Academy Music Therapy Research Centre GAMUT, Unifob Health; Brynjulf Stige, PhD, Study Director — University of Bergen/Grieg Academy Music Therapy Research Centre GAMUT, Unifob Health
Locations (5):
- Sunshine Hospital/University of Melbourne, Faculty of Music, Melbourne, Australia
- Wagner Jauregg Hospital, Linz, Austria
- Norway (3):
  - Jæren District Psychiatric Centre, Bryne, Rogaland
  - Stavanger University Hospital, Stavanger, Rogaland
  - Nordfjord Psychiatry Centre, Nordfjordeid, Sogn Og Fjordane

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolvsjord R, Gold C, Stige B. Research rigour and therapeutic flexibility: Rationale for a therapy manual developed for a randomised controlled trial. Nordic Journal of Music Therapy 14(1):15-32, 2005.
- [Background] Gold C, Rolvsjord R, Aaro LE, Aarre T, Tjemsland L, Stige B. Resource-oriented music therapy for psychiatric patients with low therapy motivation: protocol for a randomised controlled trial [NCT00137189]. BMC Psychiatry. 2005 Oct 31;5:39. doi: 10.1186/1471-244X-5-39. PMID 16259626
- [Result] Gold C, Mossler K, Grocke D, Heldal TO, Tjemsland L, Aarre T, Aaro LE, Rittmannsberger H, Stige B, Assmus J, Rolvsjord R. Individual music therapy for mental health care clients with low therapy motivation: multicentre randomised controlled trial. Psychother Psychosom. 2013;82(5):319-31. doi: 10.1159/000348452. Epub 2013 Aug 9. PMID 23942318